CLINICAL TRIAL: NCT05337904
Title: Deep Brain Stimulation: Towards a Novel Intervention Focused on the Recovery of Patients With Treatment-Resistant Schizophrenia: Randomized, Controlled, Crossover Pilot Study
Brief Title: Deep Brain Stimulation Recovery in Treatment-Resistant Schizophrenia
Acronym: DBS-R
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-ECP-2019-98
Record Dates: First submitted 2022-03-17; First posted 2022-04-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Treatment-resistant Schizophrenia; Deep Brain Stimulation
Keywords: Recovery; Deep brain stimulation; Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia

STUDY DESIGN:
Intervention Model Description: A clinical trial with four periods will be performed: pre-treatment, Intervention and follow-up, Cross-over period, and Recoveryoriented intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- On-Stimulation (Active Comparator): Disease condition is assessed with stimulation turned "on"
  Interventions: Device: On-Stimulation
- Off-Stimulation (Placebo Comparator): Disease condition is assessed with stimulation turned "off"
  Interventions: Device: Off-Stimulation

INTERVENTIONS:
Device: On-Stimulation — The surgical electrode implanted in target 1 (ACC) or target 2 (NAcc) by a pulse generating device is "on".
  Arms: On-Stimulation
Device: Off-Stimulation — The surgical electrode implanted in target 1 (ACC) or target 2 (NAcc) by a pulse generating device is "off".
  Arms: Off-Stimulation

SUMMARY:
The purpose of this project is to improve the clinical response and personal recovery of patients with treatment-resistant schizophrenia (TRS).

DETAILED DESCRIPTION:
The Project aims to improve the efficacy of the first worldwide study of Deep Brain Stimulation (DBS) carried out in our hospital -PI12 / 00042: Deep Brain Stimulation in the treatment of refractory schizophrenia- through the implementation of a white matter tractography approach, which have demonstrated to improve efficacy in other DBS studies .

Moreover, and in line with the National Strategy of Mental Health of the National Health System, this project aims to promote integrated and comprehensive care for patients with mental illness by multidisciplinary teams which includes family care, as we consider it is important to add to the DBS treatment program, a psychological intervention module based on the recovery model. Therefore, the main objectives of the present project are:

i) to optimizethe efficacy and tolerability of DBS in TRS;

ii) investigate whether the REFOCUS intervention improves the recovery of patients who are being treated with DBS. To this end, a double-blind, randomized, crossover clinical trial of DBS will be performed for 6 patients with TRS. Patients will be randomized to receive tractography-based target guidance DBS in the anterior cingulate cortex (ACC) or the nucleus accumbens (Nac). The 21 patient previously intervened with DBS (Affective disorders and TRS) and the ones included in this project, will enter into a psychological intervention phase, based on the REFOCUS model

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-50 years
* Meet DSM-5 criteria for schizophrenia, with a duration of illness < than 15 years.
* Meet updated TRS criteria.
* Non-sustained response to electroconvulsive therapy.

Exclusion Criteria:

* Contraindications to neurosurgery or DBS
* Epilepsy or seizures clozapine-induced
* Suicidal or self-harming behaviour in the last 6 months
* Other psychiatric disorders (including personality disorders)
* Significant cognitive impairment (Vocabulary test WAIS IV-TR, IQ <70, and SCIP<55)
* Severe medical non-controlled diseases
* Pregnancy or breastfeeding
* Substance use disorders (except nicotine)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Changes from baseline score to 1-3 weeks scores and to fortnightly scores until the end of trial (12 months)
  Scale to assess changes in schizophrenia' symptoms

SECONDARY OUTCOMES:
Questionnaire about the Process of Recovery (QPR) | Changes from baseline total score to 1-12 months total scores
  Scale to assess personal recovery changes
Rosenberg Self-Esteem Scale (RSES) | Changes from baseline total score to 12 months total scores
  Scale to assess a person's global self-esteem
Herth Hope Index (HHI) | Changes from baseline total score to 12 months total scores
  Scale to assess hope
Internalized stigma of mental illness scale (ISMI) | Changes from baseline total score to 12 months total scores
  Scale to assess insight
Beck Cognitive Insight Scale (BCIS) | Changes from baseline total score to 12 months total scores
  Scale to assess cognitive insight
Personal Beliefs about Illness Questionnaire-Revised (PBIQ-R) | Changes from baseline total score to 12 months total scores
  Scale to assess psychological reactions to psychosis
Trail Making Test (TMT A & B) | Changes from baseline score to 12 months score.
  Scale to assess executive function
Rey Auditory Verbal Learning Test (RAVLT) | Changes from baseline score to 12 months score.
  Scale to assess short-term auditory-verbal memory
F-A-S Test | Changes from baseline score to 12 months score.
  Scale to assess verbal fluency
Wisconsin Card Sorting Test (WCST) | Changes from baseline score to 12 months score.
  Scale to assess cognitive flexibility and abstract reasoning
Personal and Social Performance scale (PSP) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess changes in functioning
EuroQol 5 dimensions-5 levels (EQ-5D-5L) | Changes from baseline score to 1-12 months scores
  Scales to asses the patient quality of life
Client Satisfaction Questionnaire-8 (CSQ-8) | Changes from baseline score to 12 months score.
  Scales to asses the satisfaction with the treatment
Scale for the Assessment of Negative Symptoms (SANS) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scales to assess negative symptoms of schizophrenia
Clinical Global Impression - Schizophrenia (CGI-SCH) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess the severity of disorder and the degree of change in patients
Starkstein Apathy Scale (SAS) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess apathy
Beck Depression Inventory (BDI) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess depression
Beck Anxiety Inventory (BAI) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess anxiety
Global Assessment of Functioning (GAF) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to rate how serious a mental disorder may be
Side Effect Rating Scale (UKU) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to rate side effects

CONTACTS AND LOCATIONS:
Overall Officials: Iluminada Corripio, PhD, Principal Investigator — Department of Psychiatry. Hospital Santa Creu i Sant Pau
Locations (1):
- Department of Psychiatry. Hospital Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No